CLINICAL TRIAL: NCT04545138
Title: Effects of Combining Cognitive and Treadmill Training on Cognitive Function and Walking Performance-Exploration in Chronic Stroke Patient With Cognitive Impairment
Brief Title: Combining Cognitive and Treadmill Training on Cognition and Walking Performance in Stroke With Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM109069F
Record Dates: First submitted 2020-08-13; First posted 2020-09-10 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2020-07

CONDITIONS: Stroke; Cognitive Impairment
Keywords: Stroke; Cognitive Impairment; Cognitive and treadmill training
MeSH Terms: conditions — Stroke; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cognitive training during treadmill training group (Experimental): Cognitive training combine treadmill training is an intervention that can challenge participants by practicing different tasks simultaneously.
  Interventions: Other: cognitive training combine treadmill training
- treadmill training group (Active Comparator): Treadmill training as an active control.
  Interventions: Other: Treadmill training

INTERVENTIONS:
Other: cognitive training combine treadmill training — Treadmill training includes warming up for 3 minutes, training for 25 minutes, and relaxing for 2 minutes. The speed of the treadmill during the warm-up and relaxation period is based on the participant's Borg's rating of perceived exertion (RPE) 7-9 points (very slight to very slight), and the RPE during the training period does not exceed 10~12 points (slight), and ensures that patients can be cognitively trained at the same time. The cognitive training tasks will be projected on the screen and the participant have to answer the task orders during treadmill training simultaneously.
  Arms: cognitive training during treadmill training group
Other: Treadmill training — Treadmill training includes warming up for 3 minutes, training for 25 minutes, and relaxing for 2 minutes. The speed of the treadmill during the warm-up and relaxation period is based on the participant's Borg's rating of perceived exertion (RPE) 7-9 points (very slight to very slight), and the RPE during the training period does not exceed 10~12 points (slight).
  Arms: treadmill training group

SUMMARY:
Post-stroke cognitive impairment is common in stroke survivors. Cognitive function is related to walking ability. The dual task walking is required for daily activities, however, such ability is even more challenging than single walking for people with stroke. The purpose of present study is to investigate the effects of combining cognitive and treadmill training on cognitive function and dual task walking performance in chronic stroke patients with cognitive impairment.

DETAILED DESCRIPTION:
This is a single-blinded, randomized controlled trial with pre- and post-measurements. 24 subjects will be recruited, and randomly assigned to one of two groups: cognitive training during treadmill training group (experimental group) and treadmill training group (control group). The intervention for both group will be 30 minutes per session, 3 sessions per week for a total of 4 weeks. Statistical data analysis will use the SPSS 25.0. Baseline characteristics will be analyzed using independent t-test or Chi-square test. Repeated measures two-way analysis of variance (ANOVA) with Tukey's post-hoc analysis will be used to compare between time and groups. The significant level is set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* age over 50 years old
* chronic stroke (onset >6 months)
* with mini-mental state examination (MMSE) score≧24
* Montreal cognitive assessment (MoCA) score<26 (impaired cognition)
* ability to walk independently for at least 10 meters without assistive devices or support
* ability to read and write cognitive tests

Exclusion Criteria:

* diagnosis of dementia
* unstable physical condition
* any neurological, psychiatric disorder, or diagnosed with learning disability which may affect participation in this study
* visual or auditory disturbances

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2021-11-22 (Actual)

PRIMARY OUTCOMES:
Trail-making test A&B | 8 minutes
  executive function (s)
Stroop test | 10 minutes
  attention (number)
Digit span test | 8 minutes
  memory (number)
Clock drawing test | 10 minutes
  visuospatial function (score 1-10)

SECONDARY OUTCOMES:
Single walking performance- speed (cm/s) | 3 minutes
  walking speed in centimeters per second will be calculated during the single walking by using the GaitRite system
Single walking performance-step length (cm) | 3 minutes
  step length in centimeters will be calculated during the single walking by using the GaitRite system
Single walking performance-step time (s) | 3 minutes
  step time in seconds will be calculated during the single walking by using the GaitRite system
Single walking performance-cadence (steps/min) | 3 minutes
  cadence in steps per minute will be calculated during the single walking by using the GaitRite system
Cognitive dual task walking performance-speed (cm/s) | 3 minutes
  walking speed in centimeters per second will be calculated during the cognitive dual task walking by using the GaitRite system
Cognitive dual task walking performance-step length (cm) | 3 minutes
  step length in centimeters will be calculated during the cognitive dual task walking by using the GaitRite system
Cognitive dual task walking performance-step time (s) | 3 minutes
  step time in seconds will be calculated during the cognitive dual task walking by using the GaitRite system
Cognitive dual task walking performance-cadence (steps/min) | 3 minutes
  cadence in steps per minute will be calculated during the cognitive dual task walking by using the GaitRite system
Cognitive dual task walking performance-dual task cost (%) | 3 minutes
  dual task cost (%) will be calculated with the following formula: [(dual-task performance-single task performance) / single task performance] × 100%

CONTACTS AND LOCATIONS:
Overall Officials: Ray-Yau Wang, professor, Principal Investigator — National Yang Ming Chiao Tung University; Yun-Hsien Liu, Study Chair — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Beitou District, Taiwan

IPD SHARING:
Plan to Share IPD: No